CLINICAL TRIAL: NCT05006430
Title: Fecal Microbiome Changes Characterization and Safety Evaluation After Oral Administration of Lyophilized Capsules Containing Microbiota Suspension in Severe Alcoholic Hepatitis Patients: Double Blinded, Randomized, Placebo-Controlled Study.
Brief Title: Safety Evaluation of Fecal Microbiota Transplantation in Severe Alcoholic Hepatitis
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Prasun Kumar Jalal (Other)
Responsible Party: Sponsor-Investigator, Prasun Kumar Jalal, Assistant Professor of Medicine-Hepatology, Baylor College of Medicine
Organization: Baylor College of Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: H-43752
Record Dates: First submitted 2021-06-04; First posted 2021-08-16 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2024-08

CONDITIONS: Alcoholic Hepatitis
Keywords: Severe alcoholic hepatitis
MeSH Terms: conditions — Hepatitis, Alcoholic | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Arm (Active Comparator): Subjects will receive Standard of Care (SOC), based on AASLD/EASL guidelines and one dose of PRIM-DJ2727 (30 grams of stool/dose ~ 3 capsules) every day for a week followed by once weekly for 3 weeks, amounting to total 10 doses.
  PRIM-DJ2727 (microbiota suspension) is an intestinal microbial suspension prepared form stool obtained from carefully and thoroughly screened healthy human donors. It will be provided by University of Texas School of Public Health.
  Interventions: Biological: Fecal Microbiota Transplantation
- Placebo Arm (Placebo Comparator): Subjects will receive Standard of Care (SOC), based on AASLD/EASL guidelines and one dose of Placebo every day for a week followed by once weekly for 3 weeks, amounting to total 10 doses.
  Placebo will be identical to the investigational product but will not contain active PRIM-DJ2727.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Fecal Microbiota Transplantation — It's an intestinal microbial suspension prepared form stool obtained from carefully and thoroughly screened healthy human donors.
  Other Names: (PRIM-DJ2727); FMT
  Arms: Intervention Arm
Other: Placebo — Placebo will be identical to the investigational product but will not contain fecal material.
  Arms: Placebo Arm

SUMMARY:
This is a single center, randomized, parallel assignment, and double-blind placebo-controlled pilot study to characterize the intestinal microbiome in patients with severe Alcoholic Hepatitis (SAH) and evaluate the safety and the trends in improvement of diversity of intestinal microbiome following administration of lyophilized capsules containing microbiota suspension from well screened health donors. The study aims to enroll 50 patients with SAH who will be randomly assigned in 1:1 where 25 patients will be assigned to receive orally administered lyophilized PRIM-DJ2727 and Standard of Care (SOC) and the other 25 patients will be assigned to receive placebo and SOC for 4 weeks.

DETAILED DESCRIPTION:
Background:

Alcoholic hepatitis (AH) is a major public health problem in the United States, caused by chronic alcohol consumption of more than 40-60 g/day. Approximately 5 million Americans are diagnosed with AH, contributing to 5% of US annual mortality. A 28-day mortality rate had been reported in 30 to 50% of patients with AH. Steroid therapy has been the mainstay treatment of patients with severe AH for the last 50 years. Yet, such treatment hasn't clearly result in improvement of liver indices and survival rates among AH patients. Moreover, the use of prednisolone was associated with significant side effects and has several contraindications. Alternative therapeutic approaches have been explored but with lack of effectiveness. On the other side, shortage of organs and cost for liver transplantation are major barriers for liver transplantation in patients with AH.

There is a growing evidence suggesting that gut-derived bacterial endotoxins may play a role in alcohol-induced tissue injury and liver failure among heavy alcohol drinkers. This could be attributable to two factors: The first is decreased gastrointestinal motility. Ethanol can alter intestinal permeability by disrupting intercellular tight junctions and lead to GUT leak and translocation of the microbes. The second factor explain the association between microbiota and alcohol liver diseases is down-regulation of antimicrobial peptides induced by alterations in host immune responses in alcohol drinkers. One experimental study compared alcohol-sensitive mice (ASM) to alcohol-resistant mice (ARM). The study showed that ASM have reduced Bacteroidetes and increased level of Actinobacteria and Firmicutes and that performing fecal microbiota transplantation (FMT) from ARM to ASM yielded protection against Bacteroidetes depletion and against the alcohol-induced steatosis in ASM.

Over the last few years, multiple studies have shown that FMT is safe and more effective in treatment of recurrent clostridium difficile than the standard medical treatment. The successful use of FMT in recurrent C. difficile, lead to multiple exploratory studies assessing safety and efficacy of FMT in multiple diseases especially gastrointestinal disorders, including Primary Sclerosing Cholangitis (PSC), Inflammatory Bowel Diseases (IBD), Liver cirrhosis and Hepatic Encephalopathy. These studies showed that FMT was safe and showed signs of effectiveness that requires larger Randomized control trials (RCTs) to confirm these findings. A Recent study by Indian investigators showed that modulation of intestinal microbiota has shown to improve survival in patients with severe AH. However, the study had multiple limitations, including absence of randomization, limited number of biochemical parameters and prognostic scores used, use of Nasoduodenal tube to deliver FMT and the lack of detail profiling of intestinal microbiome.

Investigational Agent:

PRIM-DJ2727(microbiota suspension)is an intestinal microbial suspension prepared form stool obtained from carefully and thoroughly screened healthy human donors. PRIM-DJ2727 is prepared from a standard amount of healthy human stool mixed with 0.85%NaCI(normal saline) and 2% mannitol. Microbiota from a single donor will be screened before lyophilization and encapsulation. The lyophilized capsules given for each treatment contain bacteria from 10g Filtered stool. Placebo will be identical to the investigational product but will not contain intestinal bacteria.

This is a single center, randomized, parallel assignment, and double-blind placebo-controlled pilot study to be conducted in subjects with severe AH. Subjects with clinical diagnosis of severe alcoholic hepatitis (SAH) based on recommendation From the NIAAA Alcoholic Hepatitis Consortia criteria will be eligible.

After screening, the investigators aim to enroll 50 patients with SAH who will be randomly assigned in 1:1 where 25 patients will be assigned to receive orally administered lyophilized PRIM-DJ2727 and Standard of Care (SOC) and the other 25 patients will be assigned to receive placebo and SOC for 4 weeks.

This study is considered Pilot study due to small sample size as the investigators are using this Phase I study to assess the safety of the PRIM-DJ2727 Capsules in patients with Alcoholic hepatitis and to provide enough data to design and prepare for Phase II trial.

A formal sample size has not been calculated as this study is not powered to establish significance. This is a pilot study aimed at characterizing the intestinal microbiome in patients with severe AH and evaluate the safety and the trends in improvement of diversity of intestinal microbiome following administration of lyophilized capsules containing microbiota suspension (PRIM-DJ2727 capsules) from well screened health donors.

ELIGIBILITY:
Inclusion Criteria:

1. Any gender; male or female; aged 18- 75 years old.
2. Severe alcoholic hepatitis defined as 2.1 Onset of jaundice within prior 8 weeks. 2.2 Ongoing alcohol consumption of >40 g/day (3 drinks) in females or >60 g/day (4 drinks) in males for 6 months or more, with less than 60 days of abstinence before the onset of jaundice. 2.3 Aspartate aminotransferase >50, Aspartate aminotransferase/Alanine aminotransferase ratio > 1.5, BUT both values <400 IU/L.

2.4 Serum total bilirubin >3.0 mg/dl. 2.5 MELD score >15 and/or Maddrey DF score of ≥32.

Exclusion Criteria:

1. Non-alcoholic related liver diseases.
2. Patients with swallowing dysfunction at risk of aspiration.
3. Patients at risk for or with known anatomic or functional gastrointestinal (GI) obstruction or who have undergone major intra-abdominal surgery in the last year.
4. Patients who have undergone placement of a portosystemic shunt, infection of which may require prolonged antibiotics.
5. Patients with any congenital or acquired immunodeficiency (Other than liver disease)
6. Uncontrolled infections, sepsis, or GI bleeding.
7. Presence of cancer especially patients with skin cancer who is receiving or may receive systemic chemotherapy or immunotherapy during the study period.
8. Underlying disease that might be exacerbated by proposed treatments (e.g. HCV, HBV, HIV, TB).
9. Serum creatinine >2.5 mg/dl at presentation.
10. Pregnant and breastfeeding patients.
11. Active use drug addiction.
12. PI thinks their participation would pose a health risk e.g. patients with very severe AH with MELD score >30 or Maddrey DF > 60 or patient will be getting liver transplantation imminently.
13. Any other major illness/ condition that in the investigators judgment, will substantially increase the risk to the participant.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-01-21 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
To Assess survival in patients with severe alcoholic hepatitis receiving PRIM-DJ2727 capsules in comparison to standard of care. | [Day1 to 12 month]
  PRIM-DJ2727 is given orally at dose of 30 gm once daily for a week then, once weekly for 3 weeks
To assess the change in gut microbiome population associated with severe alcoholic hepatitis patients from baseline in study population at 4 weeks. | At [Baseline] [4 weeks]
  Microbiome will be characterized at baseline and at 4 weeks in terms of predominant genera and number of each genus population.
To assess the change in gut microbiome population associated with severe alcoholic hepatitis patients from baseline in study population at 6 months. | At [Baseline] [6 months]
  Microbiome will be characterized at baseline and at 6 months in terms of predominant genera and number of each genus population.
To assess the change in gut microbiome population associated with severe alcoholic hepatitis patients from baseline in study population at 9 months. | At [Baseline] [9 months]
  Microbiome will be characterized at baseline and at 9 months in terms of predominant genera and number of each genus population.
To assess the change in gut microbiome population associated with severe alcoholic hepatitis patients from baseline in study population at 12 months. | At [Baseline] [12months]
  Microbiome will be characterized at baseline and at 12 months in terms of predominant genera and number of each genus population.

SECONDARY OUTCOMES:
To assess change in the prognostic scores of Model for End Stage Liver Disease (MELD) from baseline in the study population at 4 weeks. | At [Baseline] [4 weeks]
  MELD score will be reported at baseline and at 4 weeks
To assess change in the prognostic scores of Model for End Stage Liver Disease (MELD) from baseline in the study population at 12 weeks. | At [Baseline] [12 weeks]
  MELD score will be reported at baseline and at 12 weeks.
To assess change in the prognostic scores of Model for End Stage Liver Disease (MELD) from baseline in the study population at 6 months. | At [Baseline] [6 months]
  MELD score will be reported at baseline and at 6 months.
To assess change in the prognostic scores of Model for End Stage Liver Disease (MELD) from baseline in the study population at 9 months. | At [Baseline] [9 months]
  MELD score will be reported at baseline and at 9 months.
To assess change in the prognostic scores of Model for End Stage Liver Disease (MELD) from baseline in the study population at 12 months. | At [Baseline] [12 months]
  MELD score will be reported at baseline and at 12 months.
To assess change in the Maddrey's Discriminant Function (Maddrey DF) from baseline in the study population at 4 weeks. | At [Baseline] [4 weeks]
  Maddery's Discriminant Function (Maddrey DF) score will be reported at baseline, and at 4 weeks.
To assess change in the Maddrey's Discriminant Function (Maddrey DF) from baseline in the study population at 12 weeks. | At [Baseline] [12 weeks]
  Maddery's Discriminant Function (Maddrey DF) score will be reported at baseline and at 12 weeks.
To assess change in the Maddrey's Discriminant Function (Maddrey DF) from baseline in the study population at 6 months. | At [Baseline] [6 month]
  Maddery's Discriminant Function (Maddrey DF) score will be reported at baseline, 6 months.
To assess change in the Maddrey's Discriminant Function (Maddrey DF) from baseline in the study population at 9 months. | At [Baseline] [ 9 month]
  Maddery's Discriminant Function (Maddrey DF) score will be reported at baseline and at 9 months.
To assess change in the Maddrey's Discriminant Function (Maddrey DF) from baseline in the study population at 12 months. | At [Baseline] [12 month]
  Maddery's Discriminant Function (Maddrey DF) score will be reported at baseline and at 12 months.
To assess change in the Lille Model from baseline in the study population at 4 weeks. | At [Baseline] [4 weeks]
  Lille score will be reported at baseline and at 4 weeks.
To assess change in the Lille Model from baseline in the study population at 12 weeks. | At [Baseline] [12 weeks]
  Lille score will be reported at baseline and at12 weeks.
To assess change in the Lille Model from baseline in the study population at 6 months. | At [Baseline] [6 month]
  Lille score will be reported at baseline and at 6 months.
To assess change in the Lille Model from baseline in the study population at 9 months. | At [Baseline] [ 9 month]
  Lille score will be reported at baseline and at 9 months.
To assess change in the Lille Model from baseline in the study population and at 12 months. | At [Baseline] [12 month]
  Lille score will be reported at baseline and at 12 months.
To assess change in the prognostic scores of Model for Glasgow Alcoholic Hepatitis Score (GAHS) from baseline in the study population at 4 weeks. | At [Baseline] [4 weeks]
  Glasgow Alcoholic Hepatitis Score (GAHS) will be reported at baseline and at 4 weeks.
To assess change in the prognostic scores of Model for Glasgow Alcoholic Hepatitis Score (GAHS) from baseline in the study population at 12 weeks. | At [Baseline] [12 weeks]
  Glasgow Alcoholic Hepatitis Score (GAHS) will be reported at baseline, and at 12 weeks.
To assess change in the prognostic scores of Model for Glasgow Alcoholic Hepatitis Score (GAHS) from baseline in the study population at 6 months. | At [Baseline] [6 month]
  Glasgow Alcoholic Hepatitis Score (GAHS) will be reported at baseline and at 6 months.
To assess change in the prognostic scores of Model for Glasgow Alcoholic Hepatitis Score (GAHS) from baseline in the study population at 9 months. | At [Baseline] [ 9 month]
  Glasgow Alcoholic Hepatitis Score (GAHS) will be reported at baseline and at 9 months.
To assess change in the prognostic scores of Model for Glasgow Alcoholic Hepatitis Score (GAHS) from baseline in the study population at 12 months. | At [Baseline] [12 month]
  Glasgow Alcoholic Hepatitis Score (GAHS) will be reported at baseline and at 12 months.

CONTACTS AND LOCATIONS:
Locations (1):
- Baylor St. Luke Medical Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided